CLINICAL TRIAL: NCT06800183
Title: Topical Application of Tartrazine for Enhanced Visualization of Subcutaneous Structures in Dermatology
Brief Title: Topical Tartrazine for Improved Skin Structure Visualization in Dermatology
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The investigators are revisiting in vitro and in vivo studies to ensure the ability to replicate the results of the original paper before proceeding to the pilot clinical study.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00469443
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Healthy; Dermoscopy; Optical Imaging
Keywords: Tartrazine; optical transparency; dermoscopy
MeSH Terms: interventions — Tartrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tartrazine Patch with 4 Doses across 3 Body Sites (Experimental): A four-chamber patch will be loaded with 0.5militer (mL) of tartrazine and applied to 1 cm diameter areas on the skin. Each chamber will deliver one of four different concentrations of a tartrazine solution-0.15 molar concentration (M), 0.3M, 0.6M, and 1.2M-on three distinct skin regions: the anterior forearm (representing thin skin), the abdomen (representing medium-thickness skin), and the back (representing thicker skin). This method ensures consistent, standardized, and simultaneous applications across all skin types and participants, reducing variability in the application process.
  Interventions: Drug: Four-Chamber Tartrazine Patch across 3 Body Sites

INTERVENTIONS:
Drug: Four-Chamber Tartrazine Patch across 3 Body Sites — This is a chamber patch comprising four increasing doses of tartrazine (0.15M, 0.3M, 0.6M, 1.2M). This will be applied on the forearm, abdomen, and back to represent different skin thicknesses.
  Other Names: FD&C Yellow 5; E102

SUMMARY:
The goal of this clinical trial is to learn if the topical application of tartrazine, an FDA-approved food dye, can help improve the transparency of the skin in healthy volunteers. The main questions it aims to answer are:

* Can topical tartrazine application allow for temporary skin transparency?
* What dose of tartrazine is required to achieve reversible skin transparency?

Participants will:

* Be given a patch test with four different doses of tartrazine
* Have these patch tests placed on the back, stomach, and forearm
* Have photographs taken every 5 minutes to see if transparency is achieved
* Be called 48 hours later to check for any side effects

DETAILED DESCRIPTION:
Optical imaging of biological tissues is limited by unwanted scattering and absorption of light, which restricts both the depth of imaging and the spatial resolution. This scattering occurs due to refractive index (RI) mismatches between different tissue components, such as the low RI of water-rich cytosol and the high RI of lipid-based structures. Current methods to reduce light scattering, such as the use of optical clearing agents (OCAs), often involve toxic chemicals or removal of tissue components, making them unsuitable for live imaging.

A recently published study in Science demonstrated that tartrazine, a commonly utilized food dye, is a potent OCA that achieves temporary optical transparency in living tissues. In rodent models, tartrazine was topically administered in a 0.6 M solution and showed reversible transparency effects and rendered their skin, muscle and connective tissues transparent while also providing high-resolution imaging down to the micrometer level without causing tissue damage. Imaging techniques such as laser speckle contrast imaging revealed clear visualization of cerebral blood vessels and internal organs, without needing to surgically remove tissue. Topical application in rodents caused minimal inflammation as affirmed by histological analysis. Additionally, the dye was rapidly cleared via urine and feces without signs of systemic toxicity, and after application, the dye can be washed out to further reduce exposure.

Compared to additional OCAs, tartrazine diffused through tissues more rapidly and required lower concentrations to achieve the desired transparency, resulting in faster visualization. Unlike conventional agents, tartrazine did not cause side effects such as tissue shrinkage or dehydration, making it a promising alternative for non-invasive imaging. These studies established that tartrazine, a strongly absorbing molecule, can reduce the RI mismatch between water and lipids, effectively minimizing light scattering and improving optical transparency.

Tartrazine, also known as FD&C Yellow No. 5, is a commonly utilized coloring agent found in food products, cosmetics, and medications with approved safety profiles across multiple regulatory bodies, including the US Food and Drug Administration (FDA), Joint Food and Agriculture Organization (FAO) and World Health Organization (WHO) Expert Committee on Food Additives (JECFA), and European Food Safety Authority (EFSA). Although tartrazine has been widely used in food and cosmetics, its clinical use for enhancing reversible skin transparency remains under-explored. The long-standing safety profile of tartrazine, in conjunction with the promising preclinical imaging modulation effects, justifies investigating its efficacy in humans.

Existing optical imaging techniques are limited by penetration depth and high scattering, particularly in vivo. This study aims to fill this gap by using tartrazine to improve visualization in human subjects. The potential benefits of this non-invasive technique for human applications are vast, particularly in dermatology, tumor imaging, and surgical planning. If successful, tartrazine could enable clearer, non-invasive imaging of tumors, vascular lesions, and other subcutaneous structures - providing real-time insights into disease progression and aiding in more accurate medical interventions. This clinical pilot study, with a primary focus on the feasibility of topical tartrazine for improving skin transparency, is built upon the promising results from rodent models and tartrazine's well-established safety profile in humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 and older
* Willingness to comply with study procedures
* Able to provide informed consent

Exclusion Criteria:

* Known allergies to tartrazine or related compounds
* Current or history of skin conditions such as eczema, psoriasis, or severe inflammatory diseases, defined as scoring ≥16 on the Eczema Area and Severity Index (EASI) or ≥10 on the Psoriasis Area Severity Index (PASI)
* Other atopic conditions such as asthma, allergic rhinitis, or hypersensitivity reactions
* Pregnancy or breastfeeding
* Use of immunosuppressive medications
* Any condition that may interfere with the safety or results of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-05-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Optical Transparency as Assessed by Total Transmittance Percentage | Up to 90 minutes
  To determine the optimal duration for maximum transparency, serial imaging will be conducted over the course of one 90 minute clinic visit (baseline, immediately post-application, and at 5-minute intervals until transparency plateaus). Imaging will be performed using non-invasive modalities. High-resolution dermoscopy will capture clear images of skin structures, and standardized high-quality photography will document the visible effects of transparency. These images will assess improvements in the resolution, depth, and overall image quality of subdermal structures, allowing the investigators to evaluate whether tartrazine significantly enhances visualization.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Sunshine, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ntziachristos V. Going deeper than microscopy: the optical imaging frontier in biology. Nat Methods. 2010 Aug;7(8):603-14. doi: 10.1038/nmeth.1483. Epub 2010 Jul 30. PMID 20676081
- [Result] Ou Z, Duh YS, Rommelfanger NJ, Keck CHC, Jiang S, Brinson K Jr, Zhao S, Schmidt EL, Wu X, Yang F, Cai B, Cui H, Qi W, Wu S, Tantry A, Roth R, Ding J, Chen X, Kaltschmidt JA, Brongersma ML, Hong G. Achieving optical transparency in live animals with absorbing molecules. Science. 2024 Sep 6;385(6713):eadm6869. doi: 10.1126/science.adm6869. Epub 2024 Sep 6. PMID 39236186